CLINICAL TRIAL: NCT01468909
Title: A Randomized Phase IIB Evaluation of Weekly Paclitaxel (NSC #673089) Plus Pazopanib (NSC #737754) Versus Weekly Paclitaxel Plus Placebo in the Treatment of Persistent or Recurrent Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Carcinoma
Brief Title: Paclitaxel With or Without Pazopanib Hydrochloride in Treating Patients With Persistent or Recurrent Ovarian Epithelial, Fallopian Tube, or Peritoneal Cavity Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2011-03635; NCI-2011-03635 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000716028; GOG-0186J; GOG-0186J (Other: NRG Oncology); GOG-0186J (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Paclitaxel; Taxes; pazopanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (paclitaxel and placebo) (Placebo Comparator): Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and placebo PO daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Placebo
- Arm II (paclitaxel and pazopanib hydrochloride) (Experimental): Patients receive paclitaxel as in arm I and pazopanib hydrochloride PO daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Drug: Pazopanib Hydrochloride

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW786034B; Votrient
  Arms: Arm II (paclitaxel and pazopanib hydrochloride)
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm I (paclitaxel and placebo)

SUMMARY:
This randomized phase II trial studies how well paclitaxel when given together with or without pazopanib hydrochloride works in treating patients with ovarian epithelial, fallopian tube, or peritoneal cavity cancer that is persistent or has come back. Drugs used in chemotherapy, such as paclitaxel work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Pazopanib hydrochloride may stop the growth of tumor cells by blocking blood flow to the tumor or by blocking some of the enzymes needed for cell growth. It is not yet known whether paclitaxel is more effective when given with or without pazopanib hydrochloride in treating ovarian epithelial, fallopian tube, and peritoneal cavity cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the progression-free survival hazard ratio of the combination of weekly paclitaxel and pazopanib (pazopanib hydrochloride) compared to weekly paclitaxel and placebo in patients with persistent or recurrent ovarian, fallopian tube, or primary peritoneal cancer.

SECONDARY OBJECTIVES:

I. To determine the frequency and severity of adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE).

II. To estimate and compare the proportion of patients responding to therapy by Response Evaluation Criteria in Solid Tumors (RECIST), cancer antigen 125 (CA125) response, the overall survival (OS), and the duration of response in each arm.

TERTIARY OBJECTIVES:

I. To explore the association between plasma cytokines and angiogenic markers and progression-free and overall survival.

II. To explore the association between single-nucleotide polymorphisms (SNPs) and progression-free and overall survival.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive paclitaxel intravenously (IV) over 1 hour on days 1, 8, and 15 and placebo orally (PO) daily on days 1-28.

ARM II: Patients receive paclitaxel as in Arm I and pazopanib hydrochloride PO daily on days 1-28.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma; histologic documentation of the original primary tumor is required via the pathology report
* Patients must have measurable disease or non-measurable (detectable) disease

  * Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be greater than or equal to 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI), or caliper measurement by clinical exam; or greater than or equal to 20 mm when measured by chest x-ray; lymph nodes must be greater than or equal to 15 mm in short axis when measured by CT or MRI
  * Non-measurable (detectable) disease in a patient is defined in this protocol as one who does not have measurable disease but has at least one of the following conditions:

    * Ascites and/or pleural effusion attributed to tumor
    * Solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST 1.1 definitions for target lesions
* Patients with measurable disease must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecology Oncology Group (GOG) protocol, if one exists; in general, this would refer to any active GOG phase III or Rare Tumor protocol for the same patient population; in addition, patients must not be eligible for the currently active phase II cytotoxic protocol in platinum resistant disease
* Patients who have received one prior regimen must have a GOG performance status of 0, 1, or 2
* Patients who have received two or three prior regimens must have a GOG performance status of 0 or 1
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy
* Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration
* Any other prior therapy directed at the malignant tumor, including chemotherapy, biological/targeted (non-cytotoxic) agents, and immunologic agents, must be discontinued at least three weeks prior to registration; chimeric or human or humanized monoclonal antibodies (including bevacizumab) or vascular endothelial growth factor (VEGF) receptor fusion proteins (including VEGF TRAP/aflibercept) must be discontinued for at least 12 weeks prior to registration
* At least 4 weeks must have elapsed since the patient underwent any major surgery (e.g., major: laparotomy, laparoscopy, thoracotomy, video-assisted thorascopic surgery [VATS]); there is no restriction on minor procedures (e.g., minor: central venous access catheter placement, ureteral stent placement or exchange, paracentesis, thoracentesis)
* Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound; this initial treatment may have included intraperitoneal therapy, consolidation, biologic/targeted (non-cytotoxic) agents (e.g., bevacizumab), or extended therapy administered after surgical or non-surgical assessment; if patients were treated with paclitaxel for their primary disease, this can have been given weekly or every 3 weeks
* Patients are allowed to receive, but are not required to receive, two additional cytotoxic regimens for management of recurrent or persistent disease, with no more than 1 non-platinum, non-taxane regimen; treatment with weekly paclitaxel for recurrent or persistent disease is NOT allowed
* Patients are allowed to receive, but are not required to receive, biologic/targeted (non-cytotoxic) therapy as part of their primary treatment regimen
* Patients must have NOT received any biologic/targeted (non-cytotoxic) therapy targeting the VEGF and/or platelet-derived growth factor (PDGF) pathways for management of recurrent or persistent disease
* For the purposes of this study, poly (ADP-ribose) polymerase (PARP) inhibitors will be considered "cytotoxic"; patients are allowed to receive, but are not required to receive, PARP inhibitors for management of primary or recurrent/persistent disease (either alone or in combination with cytotoxic chemotherapy); PARP inhibitors will NOT count as a prior regimen when given alone
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcL
* Platelets greater than or equal to 100,000/mcL
* Hemoglobin greater than or equal to 9 g/dL
* Prothrombin time (PT) such that international normalized ratio (INR) is less than or equal to 1.5 x upper limit of normal (ULN) (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin)
* Partial thromboplastin time (PTT) less than or equal to 1.5 x ULN
* Creatinine less than or equal to 1.5 x institutional ULN
* Urine protein should be screened by urinalysis; if urine protein is 2+ or higher, 24-hour urine protein should be obtained and the level must be < 1000 mg (< 1.0 g/24 hours [hrs]) for patient enrollment
* Bilirubin less than or equal to 1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 2.5 x ULN
* Subjects who have BOTH bilirubin greater than ULN and AST/ALT greater than ULN are not eligible
* Alkaline phosphatase less than or equal to 2.5 x ULN
* Patients must have normal baseline thyroid function tests (thyroid-stimulating hormone [TSH], T3, T4); a history of hypothyroidism and/or hyperthyroidism is allowed, as long as the patient has stable well-controlled thyroid function for a minimum of 2 months
* Neuropathy (sensory and motor) less than or equal to grade 1
* Patients of childbearing potential must have a negative pregnancy test prior to the study entry and be practicing an effective form of contraception; pregnant women are excluded from this study
* Patients must have signed an approved informed consent and authorization permitting the release of personal health information
* Patients must be capable of taking and absorbing oral medications; a patient must be clear of the following:

  * Any lesion, whether induced by tumor, radiation, or other conditions, which makes it difficult to swallow tablets
  * Prior surgical procedures affecting absorption including, but not limited to major resection of stomach or small bowel
  * Active peptic ulcer disease
  * Malabsorption syndrome
* Any concomitant medications that are associated with a risk of corrected QT (QTc) prolongation and/or Torsades de Pointes should be discontinued or replaced with drugs that do not carry these risks, if possible; patients who must take medication with a risk of possible risk of Torsades de Pointes should be watched carefully for symptoms of QTc prolongation, such as syncope
* Patients with personal or family history of congenital long QTc syndrome are NOT eligible
* Strong inhibitors of cytochrome P-450 system (CYP)3A4 are prohibited
* Strong inducers of CYP3A4 are prohibited
* Concomitant use of agents with narrow therapeutic windows that are metabolized by CYP3A4, CYP2D6, or CYP2C8 is not recommended

Exclusion Criteria:

* Patients who have had previous treatment with pazopanib; patients who have had previous treatment with weekly paclitaxel for recurrent or persistent disease
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis within the last three years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last three years; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients with clinically significant cardiovascular disease; this includes:

  * Uncontrolled hypertension, defined as systolic greater than 140 mm Hg or diastolic greater than 90 mm Hg despite antihypertensive medications
  * Congenital long QT syndrome or baseline QTc greater than 480 milliseconds
  * Myocardial infarction or unstable angina within 6 months prior to registration
  * New York Heart Association (NYHA) class II or greater congestive heart failure
  * History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation) or serious cardiac arrhythmia requiring medication

    * This does not include asymptomatic atrial fibrillation with controlled ventricular rate
  * Patients who have received prior treatment with an anthracycline (including doxorubicin and/or liposomal doxorubicin) must have an echocardiogram assessment and are excluded if they have an ejection fraction less than 50%
  * CTCAE grade 2 or greater peripheral vascular disease (at least brief [less than 24 hours] episodes of ischemia managed non-surgically and without permanent deficit)
  * History of cardiac angioplasty or stenting within 6 months prior to registration
  * History of coronary artery bypass graft surgery within 6 months prior to registration
  * Arterial thrombosis within 6 months prior to registration
* Patients with serious non-healing wound, ulcer, or bone fracture; this includes history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days prior to the first date of study treatment
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures which are not controlled with non-enzyme inducing anticonvulsants, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months prior to the first date of study treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pazopanib
* Known human immunodeficiency virus (HIV)-positive subjects on combination antiretroviral therapy
* Patients with any condition that may increase the risk of gastrointestinal bleeding or gastrointestinal perforation, including:

  * Active peptic ulcer disease
  * Known gastrointestinal intraluminal metastatic lesions (gastrointestinal serosa metastatic lesions are permitted)
  * Inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease)
  * Patients with clinical symptoms or signs of gastrointestinal obstruction
  * Patients who require parenteral hydration and/or nutrition
* Patients who are pregnant or nursing
* History of hemoptysis in excess of 2.5 mL (½ teaspoon) within 8 weeks prior to first dose of pazopanib
* Uncontrolled intercurrent illness including, but not limited to, psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-12-12 (Actual); Primary Completion 2018-01-27 (Actual); Study Completion 2018-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Richardson, Principal Investigator — NRG Oncology
Locations (142):
- United States (142):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Gynecologic Oncology Group of Arizona, Phoenix, Arizona
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Gynecologic Oncology Associates-Newport Beach, Newport Beach, California
  - University of Connecticut, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Florida Hospital Orlando, Orlando, Florida
  - Women's Cancer Associates, St. Petersburg, Florida
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Freeman Health System, Joplin, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Women's Cancer Care Associates LLC, Albany, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas
  - PeaceHealth Medical Group PC, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Richardson DL, Sill MW, Coleman RL, Sood AK, Pearl ML, Kehoe SM, Carney ME, Hanjani P, Van Le L, Zhou XC, Alvarez Secord A, Gray HJ, Landrum LM, Lankes HA, Hu W, Aghajanian C. Paclitaxel With and Without Pazopanib for Persistent or Recurrent Ovarian Cancer: A Randomized Clinical Trial. JAMA Oncol. 2018 Feb 1;4(2):196-202. doi: 10.1001/jamaoncol.2017.4218. PMID 29242937

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 106 patients were enrolled between December 2011 and April 2013.
Groups:
- Paclitaxel + Placebo: Paclitaxel 80 mg/m2 administered weekly on days 1, 8 and 15 with Placebo PO daily
- Paclitaxel + Pazopanib: Paclitaxel 80 mg/m2 administered weekly on days 1, 8 and 15 with Pazopanib 800 mg PO daily
Period: Overall Study
Arm/Group | Paclitaxel + Placebo | Paclitaxel + Pazopanib
Started | 52 | 54
Completed | 50 | 52
Not Completed | 2 | 2
Not completed — Never Treated | 2 | 2

BASELINE CHARACTERISTICS:
Population: All registered patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel + Placebo | Paclitaxel + Pazopanib | Total
Number analyzed (Participants) | 52 | 54 | 106
Age, Customized [Count of Participants; unit: Participants]
  Age: 30-39 years | 2 | 1 | 3
  Age: 40-49 years | 7 | 5 | 12
  Age: 50-59 years | 14 | 17 | 31
  Age: 60-69 years | 18 | 18 | 36
  Age: 70-79 years | 10 | 10 | 20
  Age: 80 + years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 54 | 106
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 4 | 7
  White | 42 | 46 | 88
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: The time from randomization until disease progression, death, or date of last contact. Endpoints are progression or death. Patients who are not observed with an endpoint are censored. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: For those patients whose disease can be evaluated by physical examination, progression was assessed prior to each 21-day cycle. CT scan or MRI if used to follow lesion for measurable disease every other cycle, Up to 5 years
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel + Placebo | Paclitaxel + Pazopanib
Number analyzed (Participants) | 52 | 54
months | 6.2 [5.5 to 8.5] | 7.5 [5.3 to 9.1]

2. Secondary Outcome: Adverse Events as Assessed by CTCAE v.4
Description: All grade 3 or greater Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported.
Time Frame: From baseline to 30 days after last dose of drug.
Population: Treated and eligible patients
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Paclitaxel + Placebo | Paclitaxel + Pazopanib
Number analyzed (Participants) | 50 | 52
participants | 18 [11 to 26] | 45 [38 to 49]

3. Secondary Outcome: Proportion of Participants With Tumor Response by RECIST
Description: Patients with Complete and Partial Tumor Response by RECIST 1.1. Responses (CR and PR) require confirmation at greater than or equal to 4 weeks from initial documentation. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Every other cycle for 6 months, then every 3 months until disease progression,Up to 5 years
Population: All randomized patients.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Paclitaxel + Placebo | Paclitaxel + Pazopanib
Number analyzed (Participants) | 52 | 54
proportion of participants | 0.192 [0.096 to 0.325] | 0.259 [0.150 to 0.397]

4. Secondary Outcome: Percentage of Participants With Tumor Response by CA-125
Description: Response as evaluated by CA-125 levels. Response is indicated if CA-125 reduced by 50% of the baseline measure.
Time Frame: Prior to each cycle of treatment. Then follow-up every three months for 2 years and then every 6 months for 3 years, up to 5 years.
Population: CA-125 Evaluable patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paclitaxel + Placebo | Paclitaxel + Pazopanib
Number analyzed (Participants) | 32 | 39
percentage of participants | 41 [24 to 59] | 72 [55 to 85]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival
Time Frame: Every cycle while patient is receiving protocol therapy. Patients monitored for survival after off therapy every 3 months for 2 years, then every 6 months, up to 5 years
Population: All randomized patients.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Paclitaxel + Placebo | Paclitaxel + Pazopanib
Number analyzed (Participants) | 52 | 54
months | 23.3 [17.3 to NA] — There are not enough deaths to determine the upper bound of the 90% confidence interval using the method provided by SAS. | 20.7 [17.0 to 22.6]

6. Other Pre Specified Outcome: Single-nucleotide Polymorphisms, Assessed Using the iPLEX Assay on the Sequenome MassARRAY Platform
Description: Analyzed using deoxyribonucleic acid isolated from whole blood specimens.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Every 28 days (1cycle) while on study treatment. Up to 30 days after treatment ends, up to 5 years.
Arm/Group | Paclitaxel + Placebo | Paclitaxel + Pazopanib
All-Cause Mortality (participants affected / at risk) | 20/50 | 23/52
Serious Adverse Events (participants affected / at risk) | 15/50 | 22/52
Other Adverse Events (participants affected / at risk) | 50/50 | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel + Placebo (N=50) | Paclitaxel + Pazopanib (N=52)
Cardiac Disorders - Other (Cardiac disorders) | 1 | 0
Optic Nerve Disorder (Eye disorders) | 0 | 1
Colonic Perforation (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Small Intestinal Perforation (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 2
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Mucositis Oral (Gastrointestinal disorders) | 0 | 1
Ileal Obstruction (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 0
Pain (General disorders) | 0 | 2
Multi-Organ Failure (General disorders) | 0 | 1
Sudden Death Nos (General disorders) | 0 | 1
Skin Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Bronchial Infection (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil Count Decreased (Investigations) | 1 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Thromboembolic Event (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel + Placebo (N=50) | Paclitaxel + Pazopanib (N=52)
Lymph Node Pain (Blood and lymphatic system disorders) | 3 | 0
Anemia (Blood and lymphatic system disorders) | 46 | 48
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 2 | 3
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1 | 0
Atrioventricular Block First Degree (Cardiac disorders) | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 3 | 2
Chest Pain - Cardiac (Cardiac disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 2
Ear Pain (Ear and labyrinth disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Eye Disorders - Other (Eye disorders) | 1 | 1
Watering Eyes (Eye disorders) | 0 | 3
Cataract (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Blurred Vision (Eye disorders) | 2 | 3
Dry Eye (Eye disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 3
Duodenal Stenosis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 6 | 4
Dry Mouth (Gastrointestinal disorders) | 2 | 4
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 27 | 23
Diarrhea (Gastrointestinal disorders) | 15 | 35
Vomiting (Gastrointestinal disorders) | 10 | 22
Bloating (Gastrointestinal disorders) | 5 | 5
Stomach Pain (Gastrointestinal disorders) | 4 | 4
Anal Hemorrhage (Gastrointestinal disorders) | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 24 | 21
Rectal Hemorrhage (Gastrointestinal disorders) | 3 | 2
Oral Dysesthesia (Gastrointestinal disorders) | 0 | 1
Mucositis Oral (Gastrointestinal disorders) | 6 | 14
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 2 | 0
Oral Hemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 2 | 0
Gingival Pain (Gastrointestinal disorders) | 0 | 1
Oral Pain (Gastrointestinal disorders) | 2 | 4
Oral Cavity Fistula (Gastrointestinal disorders) | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 30 | 36
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 4
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 3
Esophageal Stenosis (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 5
Toothache (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 2 | 3
Pain (General disorders) | 9 | 9
Malaise (General disorders) | 1 | 3
Localized Edema (General disorders) | 3 | 2
Flu Like Symptoms (General disorders) | 2 | 1
Non-Cardiac Chest Pain (General disorders) | 2 | 2
Edema Limbs (General disorders) | 7 | 8
Edema Face (General disorders) | 0 | 1
Fatigue (General disorders) | 39 | 39
Fever (General disorders) | 3 | 5
Gait Disturbance (General disorders) | 1 | 4
Chills (General disorders) | 0 | 2
Infusion Related Reaction (General disorders) | 1 | 1
Allergic Reaction (Immune system disorders) | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 3 | 4
Tooth Infection (Infections and infestations) | 1 | 0
Vulval Infection (Infections and infestations) | 0 | 1
Skin Infection (Infections and infestations) | 3 | 3
Sinusitis (Infections and infestations) | 1 | 3
Sepsis (Infections and infestations) | 1 | 0
Nail Infection (Infections and infestations) | 0 | 1
Mucosal Infection (Infections and infestations) | 1 | 1
Lung Infection (Infections and infestations) | 2 | 0
Kidney Infection (Infections and infestations) | 1 | 0
Gum Infection (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 5
Catheter Related Infection (Infections and infestations) | 1 | 1
Breast Infection (Infections and infestations) | 1 | 0
Lip Infection (Infections and infestations) | 0 | 1
Abdominal Infection (Infections and infestations) | 0 | 1
Prolapse Of Intestinal Stoma (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Wound Complication (Injury, poisoning and procedural complications) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 1
Investigations - Other (Investigations) | 1 | 0
Weight Loss (Investigations) | 1 | 6
Weight Gain (Investigations) | 2 | 3
Serum Amylase Increased (Investigations) | 1 | 0
Platelet Count Decreased (Investigations) | 10 | 24
Lymphocyte Count Decreased (Investigations) | 9 | 14
Lipase Increased (Investigations) | 1 | 1
Inr Increased (Investigations) | 2 | 1
Ggt Increased (Investigations) | 0 | 1
Electrocardiogram Qt Corrected Interval Prolonged (Investigations) | 2 | 1
Creatinine Increased (Investigations) | 5 | 10
Cholesterol High (Investigations) | 1 | 0
Neutrophil Count Decreased (Investigations) | 23 | 43
Cardiac Troponin I Increased (Investigations) | 1 | 0
Cpk Increased (Investigations) | 0 | 1
Blood Bilirubin Increased (Investigations) | 4 | 6
White Blood Cell Decreased (Investigations) | 35 | 47
Aspartate Aminotransferase Increased (Investigations) | 3 | 18
Alkaline Phosphatase Increased (Investigations) | 6 | 14
Alanine Aminotransferase Increased (Investigations) | 7 | 20
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 2
Metabolism And Nutrition Disorders - Other (Metabolism and nutrition disorders) | 0 | 1
Iron Overload (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 8
Hyponatremia (Metabolism and nutrition disorders) | 7 | 12
Hypomagnesemia (Metabolism and nutrition disorders) | 12 | 19
Hypokalemia (Metabolism and nutrition disorders) | 11 | 17
Hypoglycemia (Metabolism and nutrition disorders) | 4 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 8 | 12
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 | 12
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 3 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 17 | 21
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1
Glucose Intolerance (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 8
Anorexia (Metabolism and nutrition disorders) | 12 | 20
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 14
Muscle Weakness Trunk (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 | 6
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 10 | 11
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 8
Musculoskeletal And Connective Tissue Disorder - (Musculoskeletal and connective tissue disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 2
Transient Ischemic Attacks (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 27 | 27
Peripheral Motor Neuropathy (Nervous system disorders) | 5 | 5
Paresthesia (Nervous system disorders) | 6 | 1
Memory Impairment (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 13 | 17
Dysphasia (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 7 | 8
Dysesthesia (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 6 | 14
Concentration Impairment (Nervous system disorders) | 0 | 1
Cognitive Disturbance (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 8 | 13
Depression (Psychiatric disorders) | 3 | 9
Confusion (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 9 | 9
Urine Discoloration (Renal and urinary disorders) | 0 | 1
Urinary Urgency (Renal and urinary disorders) | 1 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 1
Urinary Incontinence (Renal and urinary disorders) | 1 | 2
Urinary Tract Pain (Renal and urinary disorders) | 2 | 2
Urinary Frequency (Renal and urinary disorders) | 1 | 1
Renal Calculi (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 4
Hematuria (Renal and urinary disorders) | 1 | 1
Cystitis Noninfective (Renal and urinary disorders) | 0 | 1
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 2
Vaginal Pain (Reproductive system and breast disorders) | 0 | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1 | 1
Pelvic Pain (Reproductive system and breast disorders) | 2 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 2
Breast Pain (Reproductive system and breast disorders) | 1 | 1
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 13
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchopulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 3
Pain Of Skin (Skin and subcutaneous tissue disorders) | 1 | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 9 | 8
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 3
Nail Ridging (Skin and subcutaneous tissue disorders) | 1 | 2
Nail Loss (Skin and subcutaneous tissue disorders) | 0 | 4
Nail Discoloration (Skin and subcutaneous tissue disorders) | 4 | 6
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 29 | 24
Surgical And Medical Procedures - Other (Surgical and medical procedures) | 0 | 1
Thromboembolic Event (Vascular disorders) | 2 | 2
Lymphedema (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 2 | 3
Hypertension (Vascular disorders) | 10 | 29
Hot Flashes (Vascular disorders) | 3 | 3
Hematoma (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT01468909/Prot_SAP_000.pdf